CLINICAL TRIAL: NCT01751282
Title: A Randomized, Double-Blind, Controlled Study to Evaluate the Effectiveness of the Use of Bone Marrow-Derived Mesenchymal Stem Cells (MSCs) in Fibrin in the Treatment of Chronic Wounds
Brief Title: Study of the Effectiveness of Autologous Bone Marrow-Derived Mesenchymal Stem Cells in Fibrin to Treat Chronic Wounds
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Left Institution where study was approved
Sponsor: Roger Williams Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: RO1AR06034201A1
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Non Healing Wounds
Keywords: Stem Cells; chronic wounds; fibrin; Bone marrow-derived mesenchymal stem cells

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard therapy and control saline spray (Placebo Comparator): Conventional standard therapy and control saline spray
  Interventions: Genetic: Stem Cell
- standard therapy and fibrin spray (Sham Comparator): Conventional standard therapy and fibrin spray
  Interventions: Genetic: Stem Cell
- Conventional standard therapy and MSCs (Experimental): Conventional Standard Therapy and MSCs (autologous bone marrow-derived mesenchymal stem cells) in fibrin spray.
  Interventions: Genetic: Stem Cell

INTERVENTIONS:
Genetic: Stem Cell

SUMMARY:
The purpose of this study is to determine the effectiveness of Autologous Bone Marrow-Derived Mesenchymal Stem Cells (MSCs) in the treatment of non-healing wounds.

DETAILED DESCRIPTION:
Sixty-six (66) subjects are planned to be enrolled into the trial. each subject's duration of participation will be 24 weeks on therapy with a 4 week post-treatment visit. A run-in phase of 2 weeks will be required prior to randomization/enrollment.

All subjects will receive appropriate and standard care for chronic wounds, including dressings, bandages, and off-loading, if required. All subjects will receive either saline, fibrin or MSCs in fibrin using an identical double-barreled syringe to keep the blind. Therefore, subjects will then be randomized to one of three groups:

1. conventional standard therapy and control saline spray
2. conventional standard therapy and fibrin spray
3. conventional standard therapy and MSCs (autologous bone marrow-derived mesenchymal stem cell)in fibrin spray

Screening Visit:

All inclusion and exclusion information will be reviewed to make sure that the subject is eligible for entry into the study. The following procedures will be performed during this two week period:

Biopsy - One (3 x 6 mm) biopsy will be taken from the edge of the wound for additional diagnostic tests and for culturing of cells. The second (3-4 mm) biopsy will be taken from the thigh for culturing of cells in the laboratory to assess the healing process. The thigh biopsy will then be excised by taking about 3/4 inch long by 1/4 inch wide margin from around it, and suturing it closed. The reason for this biopsy of the normal skin is so that it can be used to compare the healing process to the chronic wound.

Blood Sampling - Blood will be drawn for laboratory testing to assess the overall well-being, HIV, Hepatitis B & C and if the subject is a woman able to bear children, to test for pregnancy.

Wound Measurements - Wound measurements will be taken to determine the size of the wound and to assess for healing.

Randomization Visit:

If the wound has not reduced significantly in size, and the subject is still eligible for the study; he/she will be assigned to a study treatment. The decision as to which treatment he/she will receive will be determined by a process called randomization. Randomization is a mathematical process used to guarantee that each participant in the study has an equal chance of being assigned to any of the treatment options available.

The treatment groups that the subject may be assigned to are as follows:

Group #1 - Conventional Therapy and Control Saline Spray -The subject will receive conventional therapy, wound measurements, photography and observations. At the Day 1 treatment visit a double-barrel syringe system will be used to deliver topically normal saline to the wound. Up to 2 additional treatments will be applied at Weeks 3 & 6 (+ or - 2 or 3 days).

Group #2 -Conventional Therapy and Fibrin Spray - The subject will receive conventional therapy, wound measurements, photography, and observations. At the Day 1 treatment visit a double-barrel syringe system will be used to deliver topically fibrin alone to the wound. Up to 2 additional treatments will be applied at Weeks 3 & 6 (+ or - 2 or 3 days).

Group #3 - Conventional Therapy and Autologous Bone Marrow-Derived Mesenchymal Stem Cells in Fibrin Spray - The subject will receive conventional therapy, wound measurements, photography and observations. At the Day 1 treatment visit a double-barrel syringe system will be used to deliver topically autologous bone marrow-derived mesenchymal stem cells in fibrin. Up to 2 additional treatments will be applied at Weeks 3 & 6 (+ or - 2 or 3 days) if your wound is not healed.

Conventional Therapy - The subject will receive standard of care and accepted conventional therapy, regardless of which of the three groups you will be randomized in. This standard of care involves the use of dressings, bandages and protective ways to increase healing of your wound.

Bone Marrow Aspirate - Depending on the treatment group that the subject is assigned to, they will have either a bone marrow aspirate and/or sham (imitation) aspirate performed at this visit.

Day 1 Treatment Visit:

All groups will receive the study treatment that was assigned at the randomization visit. Wound measurements, clinical observations, wound dressings, adverse event reporting and photography will be performed.

Weekly Follow-up Visits (Weeks 1-24):

All groups will return weekly for conventional therapy, wound measurements, clinical observations, wound dressing changes, adverse event report, and photography. Two additional study treatments will be given at Weeks 3 & 6 (+ or - 2 or 3 days) if the wound is not healed.

Post-Treatment Follow-up Visit (Week 28):

All groups will return one month after 24 weeks of treatment for evaluation, wound measurements, and photography.

Follow-up wound Biopsies:

Participants in all three study treatment groups will be asked to have an additional biopsy of the wound edge at Week 6. This biopsy will only be taken if the wound has not healed.

ELIGIBILITY:
Inclusion Criteria:

-

A subject must meet the following conditions in order to be included in this trial:

* Male or female subjects 18 years of age or older with chronic wounds
* Wound present for at least 3 months with no evidence of healing
* Wound size must be less than or equal to 15 cm2 at randomization
* Subjects must understand and give written informed consent
* Subjects must agree to have biopsies performed as per protocol

Exclusion Criteria:

The presence of the following circumstances classifies a subject as unacceptable for inclusion in this trial:

* Evidence of active infection at the wound site or around the ulcer
* Requirement for the use of systemic corticosteroids or immuno- suppressive agents
* The subject is pregnant or breast-feeding
* The subject is known to be HIV positive
* The subject is known to be Hepatitis B or C positive
* Glycosylated hemoglobin A1C (HbA1C) is > 12%
* Poor nutritional status (albumin < 2.0 g/dL)
* The subject has a history of active, systemic malignancy
* Clinical evidence of bone exposure within the wound bed
* The subject has a history of noncompliance to medical regimens and is not considered reliable
* The subject is unable to understand the study evaluations and provide a written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Wound closure | 24 weeks

SECONDARY OUTCOMES:
Overall rate of wound healing reduction | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Falanga, MD, Principal Investigator — Roger Williams Medical Center
Locations (1):
- Roger Williams Medical Center, Providence, Rhode Island, United States